CLINICAL TRIAL: NCT02250872
Title: Effect of DPP4 Inhibitors on Cisplatin-induced Acute Kidney Injury
Brief Title: Effects of DPP4 Inhibitor on Cisplatin Induced Acute Kidney Injury
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: LG Life Sciences (Industry)
Responsible Party: Principal Investigator, Ki Young Na, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1408264002
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Cancer; Cisplatin Adverse Reaction
Keywords: Cisplatin; Nephrotoxicity; Gemigliptin; DPP4 inhibitor
MeSH Terms: conditions — Neoplasms | interventions — LC15-0444; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Gemigliptin and Cisplatin (Active Comparator): Gemigliptin 100mg daily in two divided doses for 8 days starting from one day before cisplatin-treatment
  Interventions: Drug: Gemigliptin; Drug: Cisplatin
- Control arm (Placebo Comparator): Placebo 100mg daily in two divided doses for 8 days starting from one day before cisplatin-treatment
  Interventions: Drug: Placebo; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemigliptin — Gemigliptin 100mg in 2 divided doses plus cisplatin
  Other Names: Zemiglo
  Arms: Experimental: Gemigliptin and Cisplatin
Drug: Placebo — 100mg in 2 divided doses plus cisplatin
  Other Names: Identical inert tablet to mimic gemigliptin (50mg)
  Arms: Control arm
Drug: Cisplatin — All patients will receive intravenous cisplatin

SUMMARY:
Cisplatin is a potent chemotherapeutic agent, however, its nephrotoxicity manifested by acute kidney injury (AKI) often limits applicability. Dipeptidylpeptidase-4 (DPP4) inhibitors are well known to improve glucose intolerance by augmentation of endogenous glucagon like peptide (GLP-1) and glucose-dependent insulinotropic peptide (GIP). DPP4 inhibitor also has the potential anti-apoptotic and renoprotective effect in a mouse model of cisplatin-induced AKI. This is a single-center, randomized, double-blind, parallel-group, placebo-controlled, prospective study to investigate the renoprotective effect of DPP4 inhibitor on cisplatin-induced AKI. A total 182 patients, who are scheduled to treat with cisplatin, will be recruited and randomly assigned to either Gemigliptin or placebo groups. Subjects will take study drugs for 8 days starting from one day before cisplatin treatment. Serum creatinine (Cr) and estimated glomerular filtration rate (eGFR) will be measured at 7 days after cisplatin treatment.

DETAILED DESCRIPTION:
This study will investigate possible renoprotective effects of DPP4 inhibitor on cisplatin induced acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* cancer patients treated with intravenous cisplatin
* written consent

Exclusion Criteria:

* Diabetes mellitus
* Chronic kidney disease stage IV-V (eGFR < 30ml/min/1.73m2)
* History of transplantation
* History of acute kidney injury before randomization
* Use of other nephrotoxic agents such as non steroidal anti-inflammatory drugs, aminoglycosides, colistin, vancomycin
* Receiving contrast media during last 72 hours
* Liver disease (bilirubin > 2 mg/dl, transaminase levels >2.5 times the upper limit normal)
* Active infection
* Patients with high risks of dehydration owing to poor oral intake
* High blood pressure (> 180/110 mmHg despite antihypertensive medications)
* Hypersensitivity to Gemigliptin or its excipients
* Low compliance to Gemigliptin treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-02 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury defined as any of the followings | up to 7 days
  * Increase in sCr by ≥ 0.3 mg/dl
  * Increase in sCr to ≥ 1.5 times baseline
  * Decrease in eGFR to ≥ 25%
  All subjects receive Gemigliptin or placebo at a total dose of 100mg (50mg twice a day) for 8 consecutive days, serum creatinine will be measured.

SECONDARY OUTCOMES:
delta Cr | Time Frame: up to 7 days
  Change of serum creatinine from baseline to 7 days after cisplatin treatment.
delta eGFR | up to 7 days
  Change of glomerular filtration rate calculated by the Chronic Kidney Disease Epidemiology Collaboration equations (CKD EPI) from baseline to 7 days after cisplatin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Young Na, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Katagiri D, Hamasaki Y, Doi K, Okamoto K, Negishi K, Nangaku M, Noiri E. Protection of glucagon-like peptide-1 in cisplatin-induced renal injury elucidates gut-kidney connection. J Am Soc Nephrol. 2013 Dec;24(12):2034-43. doi: 10.1681/ASN.2013020134. Epub 2013 Oct 3. PMID 24092928
- [Derived] Baek SH, Kim SH, Kim JW, Kim YJ, Lee KW, Na KY. Effects of a DPP4 inhibitor on cisplatin-induced acute kidney injury: study protocol for a randomized controlled trial. Trials. 2015 May 29;16:239. doi: 10.1186/s13063-015-0772-4. PMID 26021829
- See also: cisplatin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0015663271&QV1=CISPLATIN
- See also: gemigliptin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0911637199&QV1=GEMIGLIPTIN
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks